CLINICAL TRIAL: NCT04374435
Title: Evaluating the Efficacy of the Melanocyte Keratinocyte Transplantation Procedure in the Treatment of Vitiligo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The blistering device used for harvesting the third arm was discontinued by the manufacturer.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Anand Ganesan, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20173518
Record Dates: First submitted 2020-04-20; First posted 2020-05-05 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Vitiligo
Keywords: Vitiligo; Melanocyte; Keratinocyte; Transplantation; Procedure
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: The investigators have completed two arms of the study in sequential study design (each arm has done individually with no random assignment). An exploratory third arm was initiated but then suspended.
Masking Description: The patients were not randomly assigned, rather each arm has been done sequentially with a retrospective comparison of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- MKTP with Surgical Blade (Experimental): The investigator harvested skin from the donor site and skin from the recipient site using a surgical blade in the first arm of the study.
  Interventions: Procedure: MKTP with Surgical blade
- MKTP with Negative Pressure Instrument (Experimental): Blister grafting technique with dissociation of the cells was performed in the second arm of the study.
  Interventions: Device: MKTP with Negative Pressure Instrument
- Suction blister grafting without cell dissociation (Experimental): In this arm, transplanting the blisters without dissociation of the cells will be conducted.
  Interventions: Device: Suction blister grafting without cell dissociation

INTERVENTIONS:
Procedure: MKTP with Surgical blade — In this procedure, the donor skin will be harvested with a surgical blade and the donor skin will be dissociated
  Arms: MKTP with Surgical Blade
Device: MKTP with Negative Pressure Instrument — In this procedure, the investigator uses a negative pressure instrument to create a few blisters on the donor skin and use the blisters for grafting after cell dissociation.
  Arms: MKTP with Negative Pressure Instrument
Device: Suction blister grafting without cell dissociation — In this procedure, an automated suction blister device will be used to create micro domes and these micro domes will be used directly for grafting without dissociation.
  Arms: Suction blister grafting without cell dissociation

SUMMARY:
Vitiligo is a dermatologic disease characterized by depigmentation of the skin. While the loss of melanocytes observed in vitiligo is driven by the immune system, repigmentation of the skin that occurs during UV light treatment is driven by melanocytes that migrate out of the hair follicle and into the epidermis or the activation of stem cells within the epidermis. Unfortunately, some skin areas affected by vitiligo have very few hair follicle melanocytes and an indeterminate number of epidermal melanocytes and therefore unable to respond to light therapy.

This pilot study seeks to examine the relative efficacy of different harvesting methods for the melanocyte keratinocyte transplant procedure (MKTP) in the treatment of vitiligo.

In addition, this study will analyze the tissue of excess tissue harvested during the procedure to identify distinct cellular and molecular features of chronic vitiligo.

Patients in Dr. Ganesan's clinic at the UCI (University of California, Irvine) Department of Dermatology will be approached for participation in the study. The study will include both men and women and will not be limited by race or ethnicity. The investigators will exclude individuals less than 18 years old for the study as the investigators believe it would be difficult for these subjects to tolerate the melanocyte keratinocyte transplant procedure. Participants will be offered a melanocyte keratinocyte transplant procedure with one of the three different tissue harvesting methods (a blade, suction blister) and the method without dissociation (Cellutome).

This study has three arms:

1. MKTP with Surgical Blade
2. MKTP with Negative Pressure Instrument (suction blistering device).
3. Suction blister grafting without cell dissociation utilizing Cellutome (a device used for treating chronic burn wounds)

DETAILED DESCRIPTION:
In the first arm of the study, a normally pigmented area on the patient was anesthetized with 1% lidocaine with epinephrine. Using a surgical knife, the investigator removed a small portion of the epidermis that is unaffected by vitiligo from a small area (2cm2) on the patient's thigh to obtain donor cells. Epidermis that was harvested with the surgical knife was washed with Lactated Ringer's solution three times and then dissociated using trypsin to separate the cells into a single cell suspension. The recipient area to be grafted was ablated with an Erbium YAG(yttrium aluminum garnet)laser. Half of the dissociated single cells from the donor area (thigh)was then transplanted on to the area affected by vitiligo that the participant is interested in grafting (5 cm2 area).

The investigator then evaluated response to treatment in the transplanted areas at 1 day, 1 week, 1 month and 3 months, and 6 months by both photography and quantifying the VASI(Vitiligo Area Scoring Index) score.

VASI(Vitiligo Area Scoring Index)is the percentage of vitiligo involvement and is calculated in terms of hand units. One hand unit is approximately equivalent to 1% of the total body surface area.

In the second arm of the study, the investigator used a minimally invasive procedure (suction blister grafting) to sample the grafted skin and donor skin- this method can separate the epidermis from the dermis without inducing a scar. A normally pigmented area on the upper thigh was anesthetized with 1% lidocaine with epinephrine. Using a suction blister technique, the investigator removed a small portion of the epidermis that was unaffected by vitiligo from a small area (4 cm2 or 0.6 inch cm2) on the patient's thigh to obtain donor cells. Epidermis that was harvested was washed with Lactated Ringer's solution three times and then dissociated using trypsin to separate the cells into a single cell suspension. The recipient areas to be grafted were used to harvest epidermis using a suction blister device. Half of the dissociated single cells from the donor area (thigh) were then transplanted on to the area affected by vitiligo that the patient was interested in grafting (5 cm2 area or 0.7 inch2). The suction blister skin from the recipient sites was simultaneously dissociated into a single cell suspension. A portion of the remainder of the cells (from both the donor and recipient site) was subjected to flow sorting to quantify the populations of melanocytes and keratinocytes and to detailed molecular analysis (single-cell RNA sequencing and histology) to characterize the molecular features of chronic vitiligo. The investigator then evaluated response to treatment in the transplanted areas at 1 day, 1 week, 1 month and 3 months, and 6 months by both photography and quantifying the VASI score. This arm of the study is complete.

In the third arm of the study, the investigator uses a minimally invasive procedure (suction blister grafting without cell dissociation) to sample the grafted skin and donor skin- this method can separate the epidermis from the dermis without inducing a scar. A normally pigmented area on the upper thigh will be anesthetized with 1% lidocaine with epinephrine. Using an epidermal harvesting system which is a suction blister technique, the investigator will remove multiple small portions (about 128 blisters-1.8 mm in diameter) of the epidermis unaffected by vitiligo from a small normal area (5 cm2 ) on the patient's thigh to obtain donor cells and using a regular negative pressure instrument for removing four samples for histopathological study (two from the vitiligo area and two from the normal donor skin). The epidermis from the donor area (thigh) will then be transplanted on to the area affected by vitiligo that the patient is interested in grafting. Also, the four portions from the normal skin and the recipient site will be sent for the histopathological evaluation.

The investigator will then evaluate response to treatment in the transplanted areas at 1 day, 1 week, 1 month and 3 months, and 6 months by both photography, quantifying the change in depigmented surface area, and the VASI(Vitiligo Area Scoring Index) score. Also, the investigator will evaluate the two vitiligo samples and two normal skin samples through histopathology to assess where the unique populations of cells identified in their RNA-sequencing analysis are localized (obtained from arm 2). The investigator hypothesizes that his transplant procedure will yield excellent to good repigmentation, resulting in a mean of 60% reduction in surface area (SD=30%) from baseline to 6-month follow up. With a sample size of 5 patients, this study will achieve 90% power to test this hypothesis based on a two-sided paired t-test at p=0.05 significance level. In addition, the investigator will compare the results from the 7 patients harvested using the surgical blade technique (procedure already completed and follow up results pending) with the results from 7 patients harvested with the suction blisters (completed) and seven patients from the newly proposed experimental group (three completed to date).

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of vitiligo by a board-certified dermatologist
* Candidate for vitiligo treatment as determined by lead researcher
* Has a 5 cm2 area of vitiligo and an area on the upper thigh that is not affected by the disease
* Over 18 years of age at the time of signing the informed consent form
* Ability to understand, abide by and participate in study procedures

Exclusion Criteria:

* Inability to understand or abide by instructions for participation in study and procedure
* Pregnant or lactating women
* Less than 18 years old at the time of signing the informed consent form
* Current use of tobacco products or within 1 month prior to procedure date
* History of coagulation disorder, platelet dysfunction disorder, platelet count less than <150,000 platelets per microliter
* History of poor wound healing or condition that would compromise optimal healing of graft site as deemed by lead researcher
* History of keloids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand K Ganesan, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shiu J, Zhang L, Lentsch G, Flesher JL, Jin S, Polleys C, Jo SJ, Mizzoni C, Mobasher P, Kwan J, Rius-Diaz F, Tromberg BJ, Georgakoudi I, Nie Q, Balu M, Ganesan AK. Multimodal analyses of vitiligo skin identify tissue characteristics of stable disease. JCI Insight. 2022 Jul 8;7(13):e154585. doi: 10.1172/jci.insight.154585. PMID 35653192
- [Result] Mobasher P, Shiu J, Lentsch G, Ganesan AK. Comparing the Efficacy of 2 Different Harvesting Techniques for Melanocyte Keratinocyte Transplantation in Vitiligo. Dermatol Surg. 2021 May 1;47(5):732-733. doi: 10.1097/DSS.0000000000002922. No abstract available. PMID 33905400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
Started | 7 | 7 | 3
Completed | 7 | 7 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation | Total
Number analyzed (Participants) | 7 | 7 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 1 | 12
  >=65 years | 1 | 2 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 47 [26 to 79] | 51 [29 to 68] | 52 [19 to 70] | 49 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 11
  Male | 4 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 1 | 11
  Unknown or Not Reported | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 0 | 0 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had a Percent Change in Body Surface Area in Response Rate to Treatment
Description: Number of patients who had a percent change in body surface area in response rate to treatment as assessed by photography.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
Number analyzed (Participants) | 7 | 7 | 3
Participants | 6 | 4 | 2

2. Primary Outcome: Change in VASI
Description: Percent change in the transplanted areas as evaluated by VASI (Vitiligo Area Scoring Index). The negative scores mean improvement and positive scores means worsening.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in vitiligo surface area
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
Number analyzed (Participants) | 7 | 7 | 3
% change in vitiligo surface area | -23.0 (24.0) | -10.2 (18.9) | -0.33 (0.35)

3. Secondary Outcome: Percent of Patients That Healed in One Week
Description: The investigator will evaluate what percentage of patients healed at both the donor and graft site at one week.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
Number analyzed (Participants) | 7 | 7 | 3
Participants | 7 | 7 | 3

4. Secondary Outcome: Percentage of Patients That Experience Complications
Description: The investigator will record the percentage of patients that had complications in each group at either the donor or recipient site.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
Number analyzed (Participants) | 7 | 7 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MKTP With Surgical Blade | MKTP With Negative Pressure Instrument | Suction Blister Grafting Without Cell Dissociation
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT04374435/Prot_SAP_ICF_003.pdf